CLINICAL TRIAL: NCT06064526
Title: Real-world Experience of Dupilumab for the Treatment of Severe Asthma in the United Kingdom: a Retrospective Study
Brief Title: An Observational, Retrospective Multicentre Medical Record Review to Describe the Post-authorisation Early Clinical Experience of Dupilumab in the Treatment of Adult Severe Asthma
Acronym: DUPIAZA
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: CEF0101; U1111-1294-7718 (Registry Identifier: ICTRP); CEF0101 (Other: Sanofi Identifier)
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: The source population for this study is adult participants with severe asthma treated with dupilumab in routine clinical practice in the UK.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Non-interventional study based on secondary use of hospital medical records

SUMMARY:
The purpose of this retrospective medical record review is to describe the real-world clinical effectiveness of dupilumab with patients in the United Kingdom with severe asthma.

DETAILED DESCRIPTION:
Participants initiating treatment with dupilumab in the UK between 5th July 2019 and 12th August 2021 will be included in the study record review, permitting participation in research and if medical records are available for review. No intervention will be administered in this clinical trial. Data will be collected from hospital medical records and other hospital databases.

ELIGIBILITY:
Inclusion Criteria:

• Adult participants (aged ≥18 years at index) with severe asthma, initiated with dupilumab treatment (≥1 dose) between 07/05/2019 (EU licence) and 08/12/2021 • Participants with ≥1 routine asthma clinic visit recorded within 6 months prior to or on the date of dupilumab initiation and ≥1 routine asthma clinic visit recorded between 9 and 16 months post-dupilumab initiation

Exclusion Criteria:

• Participants known to have opted out of participation in research • Participants whose medical records are not available for review The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with severe asthma treated with dupilumab in routine clinical practice from medical records of nine participating centres meeting the study eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Oral corticosteroid (OCS) dose | Up to 25 months
  Measured per day
Annual asthma exacerbation rate | Up to 25 months
  The annual exacerbation rate will be calculated as the sum of OCS exacerbations and the hospital asthma exacerbations that occurred more than 7 days separated from other exacerbations. Exacerbations will be defined according to whether or not the patient was receiving asthma maintenance OCS.
Forced expiratory volume in one second (FEV1) | Up to 25 months
  FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer measured in L
Peak expiratory flow rate (PEF) | Up to 25 months
  The PEF is a participant's maximum speed of expiration, as measured with a peak flow meter measured in L/min.
Asthma Control Questionnaire (ACQ) score | Up to 25 months
  Total scores for the different versions of ACQ (5/6/7) are highly correlated and measurement properties are reported to be similar but results will be reported separately according to the version used. Differences in ACQ will only be calculated where the same version was used for the time points being compared. The score ranges from 0 (totally controlled) and 6 (severely uncontrolled). A high score indicates low asthma control.
Asthma Quality of Life Questionnaire (AQLQ) score | Up to 25 months
  Overall scores for the mini-AQLQ and the AQLQ have been reported to be very similar but results will be reported separately according to the version used. Differences in AQLQ will only be calculated where the same version was used for the time points being compared. The overall score is 1 to 7. Higher AQLQ scores indicate better health-related quality of life.

SECONDARY OUTCOMES:
Body mass index (BMI [kg/m2]) | At baseline
  Calculated as weight at baseline (kg) divided by height in m2
Inhaled corticosteroid dose | At baseline
  Measured per day
Dupilumab treatment duration | Up to 25 months
  Time from the first dose to the last recorded dose (information on treatment interruptions will not be collected).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, France, Chilly-Mazarin, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org